CLINICAL TRIAL: NCT02533544
Title: Treatment Efficacy and Safety of Tenofovir Disoproxil Fumarate (TDF) in naïve Chronic Hepatitis B : a Real Life Multicenter Cohort Study in Korea
Brief Title: Treatment Efficacy and Safety of Tenofovir Disoproxil Fumarate (TDF) in naïve Chronic Hepatitis B
Status: Completed | Type: Observational
Sponsor: Myeong Jun Song (Other)
Collaborators: Gilead Sciences (Industry); Wonkwang University (Other); Soonchunhyang University Hospital (Other); Chungnam National University Hospital (Other); Konyang University Hospital (Other)
Responsible Party: Sponsor-Investigator, Myeong Jun Song, Assistant Professor, The Catholic University of Korea
Organization: The Catholic University of Korea (Other)
Other Study IDs: IN-US-174-1805
Record Dates: First submitted 2015-08-17; First posted 2015-08-27 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Chronic Hepatitis B
Keywords: tenofovir disoproxil fumarate
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Tenofovir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- tenofovir disoproxil fumarate monotherapy: a group which treated with tenofovir disoproxil fumarate
  Interventions: Drug: tenofovir disoproxil fumarate

INTERVENTIONS:
Drug: tenofovir disoproxil fumarate

SUMMARY:
This is an open-label, single arm cohort study to see efficacy and safety of tenofovir disoproxil fumarate (TDF) in naïve chronic hepatitis B, retrospectively and prospectively both.

ELIGIBILITY:
Inclusion Criteria:

1. Must have the ability to understand and sign a written informed consent form, which must be obtained prior to initiation of study procedures.
2. Adult male and non-pregnant, non-lactating female subjects, 19 years of age and older, based on the date of the screening visit. A negative serum pregnancy test at Screening is required for female subjects of childbearing potential (unless surgically sterile or greater than 2 years post-menopausal).
3. Documented evidence of chronic HBV infection (e.g. HBsAg positive for more than 6 months)
4. Chronic hepatitis B with the following:

   * HBeAg-positive and HBeAb negative at Screening
   * Screening HBV DNA ≥ 1x 105 copies/mL
   * Screening serum ALT level ≥ ×ULN(80 IU/L) and ≤ 10 ×ULN (by center laboratory range) OR
   * HBeAg-negative and HBeAb positive at Screening
   * Screening HBV DNA ≥ 1x 104 copies/mL
   * Screening serum ALT level ≥ ×ULN(80 IU/L) and ≤ 10 ×ULN (by center laboratory range) OR
   * Cirrhosis at Screening
   * Screening HBV DNA ≥ 1x 104 copies/mL in HBeAg negative or
   * Screening HBV DNA ≥ 1x 105 copies/mL in HBeAg positive
   * Screening serum ALT level ≥ ×ULN and ≤ 10 ×ULN (by center laboratory range)
5. A patient who treating with TDF as a treatment-naïve for Hepatitis B. Treatment naïve subjects defined as no history of antiviral therapy or < 12 weeks of oral antiviral treatment with any nucleoside or nucleotide analogue, including lamivudine or adefovir, clevudine, telbivudine, entecavir
6. Decompensated liver cirrhosis defined based on a Child-Turcotte-Pugh (CTP) score ≥ 7 (Child B and C) or presence with at least one episode of ascites, jaundice, hepatic encephalopathy or variceal bleeding
7. Any previous treatment with interferon (pegylated or non-pegylated) must have ended at least 6 months prior to the baseline visit
8. Must be willing and able to comply with all study requirements.

Exclusion Criteria:

Subjects who meet any of the following exclusion criteria are not to be enrolled in the study.

1. Pregnant women, women who are breastfeeding or who believe they may wish to become pregnant during the course of the study.
2. Co-infection with HCV, HIV
3. Evidence of hepatocellular carcinoma (e.g. α-fetoprotein> 50 ng/mL or as evidenced by recent ultrasound or other standard of care measure)
4. Malignancy within 5 years prior to screening, with the exception of specific cancers that are cured by surgical resection (basal cell skin cancer, etc). Subjects under evaluation for possible malignancy are not eligible
5. Current alcohol or substance abuse judged by the investigator to potentially interfere with subject compliance
6. Currently receiving therapy with cytotoxic agent, nephrotoxic agents, or agents capable of modifying renal excretion
7. Any other clinical condition or prior therapy that, in the opinion of the Investigator, would make the subject unsuitable for the study or unable to comply with dosing requirements.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Secondary and Tertiary hospital
Sampling Method: Probability Sample
Enrollment: 572 (Actual)
Dates: Start 2015-10; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects with plasma HBV DNA levels below 116 copies/mL at Week 48 | week 48
  proportion of subjects with plasma HBV DNA levels below 116 copies/mL at Week 48
The proportion of subjects with plasma HBV DNA levels below 116 copies/mL at Week 96 | Week 96
  proportion of subjects with plasma HBV DNA levels below 116 copies/mL at Week 96

SECONDARY OUTCOMES:
The proportion of subjects with plasma HBV DNA levels below 116 copies/mL at every visits | week 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144
  The proportion of subjects with plasma HBV DNA levels below 116 copies/mL at every visits
The proportion of the biochemical (alanine aminotransferase normalization) response of TDF for the treatment of chronic hepatitis B at Week 48 and 96 | Week 48 and 96
  The proportion of the biochemical (alanine aminotransferase normalization) response of TDF for the treatment of chronic hepatitis B at Week 48 and 96
The proportion of the serological response (loss of HBeAg and seroconversion to HBeAb) of TDF for the treatment of chronic hepatitis B at Week 48 and 96 | Week 48 and 96
  The proportion of the serological response (loss of HBeAg and seroconversion to HBeAb) of TDF for the treatment of chronic hepatitis B at Week 48 and 96
The proportion of the serological response (loss of HBsAg and seroconversion to HBsAb) of TDF for the treatment of chronic hepatitis B at Week 48 and 96 | Week 48 and 96
  The proportion of the serological response (loss of HBsAg and seroconversion to HBsAb) of TDF for the treatment of chronic hepatitis B at Week 48 and 96
The change from baseline in the decline of HBV DNA at every visits | week 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144
  The change from baseline in the decline of HBV DNA at every visits
The proportion of patients showing virological breakthrough at week 48 and 96 | Week 48 and 96
  The proportion of patients showing virological breakthrough at week 48 and 96.
  Virological Breakthrough defined as any increase in serum HBV DNA by >1 log10 from nadir or redetection of serum HBV DNA at levels ≥10-fold the lower limit of detection of the HBV DNA assay after having an undetectable result
The incidence of resistance of TDF among patients showing virological breakthrough at week 48 and 96 | Week 48 and 96
  The incidence of resistance of TDF among patients showing virological breakthrough at week 48 and 96.
  Virological Breakthrough defined as any increase in serum HBV DNA by >1 log10 from nadir or redetection of serum HBV DNA at levels ≥10-fold the lower limit of detection of the HBV DNA assay after having an undetectable result
The proportion of improvement of liver function including Child Score, Model for End-stage Liver Disease (MELD) score at Week 48 and 96 | Week 48 and 96
  The proportion of improvement of liver function including Child Score, MELD score at Week 48 and 96
The proportion of improvement of Fibrosis marker including Aspartate aminotransferase to Platelet Ratio Index(APRI) at Week 48 and 96 | Week 48 and 96
  The proportion of improvement of Fibrosis marker including Aspartate aminotransferase to Platelet Ratio Index(APRI) at Week 48 and 96

CONTACTS AND LOCATIONS:
Overall Officials: Myeong Jun Song, Ph.D. M.D., Principal Investigator — The Catholic University of Korea
Locations (1):
- The Catholic University of Korea, Daejeon St.Mary's Hosptial, Junggu, Daejeon, South Korea

REFERENCES:
- [Derived] Kwon JH, Song MJ, Jang JW, Bae SH, Choi JY, Yoon SK, Kim HY, Kim CW, Song DS, Chang UI, Yang JM, You CR, Choi SW, Lee HL, Lee SW, Han NI, Nam SW, Kim SG, Kim YS, Kim SH, Lee BS, Lee TH, Cho EY. Efficacy and Safety of Tenofovir Disoproxil Fumarate in Treatment-Naive Patients with Chronic Hepatitis B in Korea. Dig Dis Sci. 2019 Jul;64(7):2039-2048. doi: 10.1007/s10620-019-05489-7. Epub 2019 Feb 6. PMID 30725293